CLINICAL TRIAL: NCT01007266
Title: Partners for Better Health in Adolescent Type 2 Diabetes: The Buddy Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100002; 10-DK-0002
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-04-14

CONDITIONS: Obesity; Diabetes Mellitus, Type 2; Abnormal Glucose Metabolism; Type 2 Diabetes
Keywords: Type 2 Diabetes Mellitus; Adolescents; Pediatric; Patient Partner; Buddy; Obesity; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

ARMS (2):
- Group A (Other): Buddy Group - Individuals with type 2 diabetes receive conventional diabetes treatment and are assigned a patient partner (Buddy)
  Interventions: Behavioral: Assignment of a Lay Patient Partner
- Group B (Active Comparator): Individuals receive conventional treatment for type 2 diabetes
  Interventions: Behavioral: Assignment of a Lay Patient Partner

INTERVENTIONS:
Behavioral: Assignment of a Lay Patient Partner

SUMMARY:
Background:

* Type 2 diabetes mellitus (T2DM) is becoming more common among youth, particularly in minority populations. Few drug treatments are approved for T2DM in adolescents, and behavioral and lifestyle factors may contribute to their difficulties in following strict treatment regimens.
* It is unknown whether a minimally invasive patient partner ( buddy ) program, which has been developed to help improve diabetes control and quality of life, will be successful in a population of pediatric patients with T2DM.

Objectives:

* To evaluate the effect of a minimally invasive intervention (being assigned a patient partner, or buddy ) on blood sugar levels in adolescents with T2DM.
* To assess changes between groups in body weight, number of home glucose monitor checks, compliance with medications, adherence to visit schedule, and psychological well-being.

Eligibility:

- Adolescents and young adults between 12 and 20 years of age who have been diagnosed with type 2 diabetes and whose blood glucose control needs improvement.

Design:

* Participants will be divided by chance into two groups: in one group, participants will have a buddy and receive standard care; while in the other group, participants will receive standard care alone.
* The buddy is not a health care professional and is not authorized to provide any medical advice.
* Participants will be followed in the study for a total of 6 months. All study participants will receive standard treatment for T2DM.
* All patients will be asked to fill out a screening questionnaire (on paper or online) at the beginning of the study and a quality of life and eating behaviors questionnaire at the beginning and at the end of the study. These forms will include questions on medical history, emotions, well-being, and eating habits.
* Participants in both groups will have one diabetes clinic visit at the NIH Clinical Center or at Children s National Medical Center (CNMC) at the beginning of the study and two follow-up visits at the NIH or CNMC approximately 3 months apart. All visits include a physical examination, detailed medical history, and laboratory testing which is part of routine care for diabetes.
* Participants assigned to the buddy group will receive phone or online messages from the buddy once a week and will meet with the buddy once a month for less than 1 hour. The purpose of the in-person visit is to get to know each other better outside the usual hospital or clinic environment. The visits should take place at home, but may also take place elsewhere, for example, at schools, cafes, or libraries chosen by both the participant and the buddy. These face-to-face meetings may also take place at NIH or at CNMC if this is more convenient.

DETAILED DESCRIPTION:
Background

Type 2 diabetes mellitus (T2DM) is becoming increasingly prevalent among youth, particularly in minority populations. Few pharmacologic agents are approved for the treatment of T2DM in adolescents, and behavioral and lifestyle factors may contribute to adolescents difficulty adhering to treatment regimens. A minimally-invasive buddy-intervention (to help improve diabetes control and to foster improvement in quality of life) has not been systematically evaluated in a population of pediatric patients with T2DM.

Objectives

1. To evaluate the effect of a minimally invasive intervention the buddy on hemoglobin A1c (HbA1c) levels in adolescents with T2DM.
2. To assess changes between groups in body weight, number of home glucose monitor checks, compliance with medications, adherence to visit schedule, and psychological well-being.

Methods

Patients will be randomized to conventional treatment versus interventional group (buddy arm), and will be followed for 6 months. During this period, all patients should undergo two visits including laboratory testing (HbA1c) approximately 3 months apart. Those in the buddy arm will have weekly phone or online contact and once-monthly home visits from the buddy (a volunteer patient partner), with the use of systematic questionnaires and a secure database for data collection and maintenance.

ELIGIBILITY:
* INCLUSION CRITERIA:

Any patient with type 2 diabetes mellitus as documented by his or her primary physician

1. Age 12-20 years at enrollment
2. Most recent HbA1c greater than or equal to 7%

EXCLUSION CRITERIA:

1. Significant comorbidity that, in the opinion of the investigators, may limit adequate study participation
2. Significant psychiatric or cognitive disorder, or communication difficulty that will, in the opinion of the investigators, limit the subject's ability to interact with the patient assistant or may present a danger to the patient assistant; patients with current suicidal or homicidal ideation, history of arrest for violent behavior, or history of school suspension/expulsion for violent behavior will be excluded.
3. Pregnancy or intention to become pregnant within 6 months

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2009-10-09; Study Completion 2013-01-24 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of a minimally invasive intervention (the buddy system) on hemoglobin A1c levels in adolescents with T2DM. | 6 months

SECONDARY OUTCOMES:
To assess changes between groups in body weight, number of home glucose monitor checks, compliance with medications, adherence to visit schedule, and psychological well-being. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kristina I Rother, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (2):
- United States (2):
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Yokoyama H, Okudaira M, Otani T, Takaike H, Miura J, Saeki A, Uchigata Y, Omori Y. Existence of early-onset NIDDM Japanese demonstrating severe diabetic complications. Diabetes Care. 1997 May;20(5):844-7. doi: 10.2337/diacare.20.5.844. PMID 9135953
- [Background] Krieger J, Collier C, Song L, Martin D. Linking community-based blood pressure measurement to clinical care: a randomized controlled trial of outreach and tracking by community health workers. Am J Public Health. 1999 Jun;89(6):856-61. doi: 10.2105/ajph.89.6.856. PMID 10358675
- [Background] Duncan GE. Prevalence of diabetes and impaired fasting glucose levels among US adolescents: National Health and Nutrition Examination Survey, 1999-2002. Arch Pediatr Adolesc Med. 2006 May;160(5):523-8. doi: 10.1001/archpedi.160.5.523. PMID 16651496